CLINICAL TRIAL: NCT01133561
Title: The CLINICAL And MOLECULAR EFFECTS Of An INSULIN SENSITIZING DRUG: 'PIOGLITAZONE'On PSORIASIS TREATMENT
Brief Title: Pioglitazone in Psoriasis- A Clinical and Molecular Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Vanessa Galal Hafez/ Assistant lecturer of Dermatology, Dermatology department, Faculty of medicine, Cairo university
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VHafez 2010
Record Dates: First submitted 2010-05-25; First posted 2010-05-31 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Psoriasis
Keywords: psoriasis; insulin resistance; metabolic syndrome; pioglitazone; randomized control trial
MeSH Terms: conditions — Psoriasis; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- actozone A (Active Comparator): Pioglitazone 30 mg tablets daily
  Interventions: Drug: actozone A
- actozone B (Placebo Comparator): placebo
  Interventions: Drug: actozone B

INTERVENTIONS:
Drug: actozone A — pioglitazone 30 mg tablet , once daily dose for 10 weeks
  Arms: actozone A
Drug: actozone B — one tablet of vehicle without active ingredient pioglitazone
  Arms: actozone B

SUMMARY:
The study will assess the effectiveness of Pioglitazone on cellular and clinical levels in terms of improvement of both skin and systemic manifestations of psoriasis.

The investigators assume that pioglitazone (one of thiazolidinediones readily available in Egypt), can regulate keratinocytes' disordered proliferation observed in psoriasis, in addition to improving the insulin resistance in peripheral tissues observed in many psoriatic patients and causing metabolic syndrome. This will allow to give a safer therapy than the available ones for psoriasis and to treat the patient in a more global perspective.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and less than 65 years.
* Plaque psoriasis vulgaris ≥ 10% (apart from palmoplantar psoriasis which will be included).

Exclusion Criteria:

* Age less than 18 years and more than 65 years
* Mild psoriasis less than 10% body surface area
* Erythrodermic or pustular psoriasis
* Liver disease, cardiac disease (suspected from history or ECG), or any other major medical disorder detected by history.
* Pregnant and lactating females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Treatment success detected as clinical improvement of skin condition | 10 weeks
  PASI improvement by at least 50% from baseline before treatment(Psoriasis Area and Severity Index)= PASI-50

SECONDARY OUTCOMES:
Fasting serum insulin reduction from baseline before treatment | 10 weeks
C-reactive protein titre reduction from baseline value before treatment | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manal AW Bosseila, MD, Study Chair — Cairo University-Dermatology department; Mona RE Abdel Halim, MD, Study Director — Cairo university- Dermatology department; Mohamed I Sheta, MD, Study Director — Cairo university- Internal medicine department; Olfat G Shaker, MD, Study Director — Cairo University- Biochemistry department
Locations (1):
- Dermatology department of cairo university faculty of medicine, Cairo, Egypt